CLINICAL TRIAL: NCT06281106
Title: Tyrosine Kinase 2 (TYK2) Inhibition in Paradoxical Psoriasis A Randomized, Double-blind, Placebo-controlled Multi-center Study Evaluating the Effect of Deucravacitinib on Severity of Psoriasis in Patients With Paradoxical Psoriasis
Brief Title: TYK2 Inhibition in Paradoxical Psoriasis
Acronym: TYPP
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: External research funds were canceled, so study could unforunately not be continued
Sponsor: Prof Curdin Conrad (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor-Investigator, Prof Curdin Conrad, Associate Professor, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM011-1118; KOFAM 2023-01731 (Other: CER-VD)
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Psoriasis
Keywords: Drug-induced Psoriasis; anti-TNF treatment; Psoriasis; Tumor necrosis factor inhibitors; Paradoxical Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib

STUDY DESIGN:
Intervention Model Description: During 4 weeks the patients of the 2 arms receive either Deucravacitinib 6mg 1x/day or an identically looking placebo.
  At Week 4, Patients with underlying disease of Crohn's disease, colitis ulcerosa, uveitis will stop the study, to avoid that they are too long without efficient treatment for their underlying disease.
  Patients with underlying disease of psoriasis or psoriatic arthritis will have the possiblity to continue in Part 2, where they all will receive Deucravacitinib 6mg 1x/day, open label for 3 months
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Lab personnel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 'Deucravacitinib' (Active Comparator): Deucravacitinib 6mg oral intake once daily for 4 weeks
  Interventions: Drug: Deucravacitinib
- 'Placebo' (Placebo Comparator): Matching Placebo oral intake once daily for 4 weeks
  Interventions: Drug: Deucravacitinib

INTERVENTIONS:
Drug: Deucravacitinib — Daily drug intake for 4 weeks.

SUMMARY:
Paradoxical psoriasis is a side effect of a biological treatment (anti-tumor necrosis factor agent, short called anti-TNF) that is used to treat diseases of the skin, the intestine or the joints. If paradoxical psoriasis occurs, the anti-TNF-treatment often needs to be stopped and so far, no specific treatment for paradoxical psoriasis exists.

This research project aims to study whether the efficacy of the drug 'Deucravacitinib' 6mg, a tablet taken by mouth once a day is superior compared to taking a placebo in treating paradoxical psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Paradoxical Psoriasis caused by anti-TNF treatment, with with Investigator Global Assessment ≥ 2 and Body Surface Area ≥ 2%
2. Females who are of child-bearing potential should be practicing highly-effective contraception methods throughout the study and for 28 days after the last dose of study drug;
3. Male subjects with a mechanical contraceptive method;
4. be in good health
5. be willing to have skin biopsies taken

Exclusion Criteria:

1. Use of any other anti-psoriatic therapy. Certain washout periods of treatments needs to be respected
2. Infection(s) requiring treatment with intravenous (IV) anti-infectives within 30 days prior to the Baseline visit or oral anti-infectives within 14 days prior to the Baseline visit;
3. A positive serology test for hepatitis B, hepatitis C, HIV;
4. History of lymphoproliferative disease or of malignancy within the past 5 years.
5. Chronic recurring bacterial infections or active tuberculosis;
6. Positive pregnancy test at Screening and at the Baseline visit;
7. Female subjects who are pregnant or breast-feeding or considering becoming pregnant during the study;
8. History of clinically significant alcohol or drug abuse in the last 12 months
9. Known hypersensitivity to Deucravacitinib or any of its excipients
10. Current severe progressive or uncontrolled disease
11. Live vaccine within 12 weeks before Baseline Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Paradoxical Psoriasis Investigator Global Assessment | At Week 4
  Percentage of patients attaining PxP IGA 0/1 and at least a reduction of 2 points from baseline

SECONDARY OUTCOMES:
Paradoxical Psoriasis Body Surface Area | At Week 4
  Change of Paradoxical Psoriasis Body Surface Area ( PxP-BSA ) measured in percentage of the total Body Surface area. 100% would be the total Body Surface area.
Paradoxical Psoriasis palmoplantar Psoriasis Area and Severity Index | at 4 Weeks
  Change of Paradoxical Psoriasis palmoplantar Psoriasis Area and Severity Index (PxP PPPASI) Score in patients presenting paradoxical psoriasis of the hands of feet. Where 72 is the worst possible calculated score, and 0 is the best score.
Paradoxical Psoriasis Scalp Investigator General Assessment | At Week 4
  Change of Paradoxical Psoriasis Scalp Investigator General Assessment (PxP-scalp IGA) if paradoxical Psoriasis is affecting the Scalp. It's a 4-point Scale with 4 being the worst score (severe Scalp Psoriasis) and 0 is the best score with clear scalp.
Psoriasis Area and Severity Index (PASI) | At Week 4 and at Week 16
  Change of Psoriasis Area and Severity Index (PASI) in patients with pre-existing disease of Psoriasis. The PASI is calculated following the official PASI Score calculation. 72 is the worst score, 0 means clear skin.
American College of Rheumatology (ACR) Score | At Week 4 and Week 16
  Percentage of patients with underlying disease of psoriasic arthritis, having an American College of Rheumatology (ACR) Score of 20%, 50% or 70% reduction in comparison with the Baseline assessment. To achive a 70% ACR, an improvement of 70% in the number of painful joints, and in the number of swollen joints must be reached, additionally an improvement of 70% in 3 out of 5 criteria need to be reached:
  Health Assessment Questionnaire, assessing patients disability (0 best score, 3 worst score), Patient overall disease assessement (0 no disease activity, 10 worst disease activity), Visual Analogue Scale assessing patients pain (0 no pain, 10 worst pain), C-reactive protein Blood-Test (CRP); Investigator General Disease Activity Assessment (0 no disease activity, 10 worst disease activity)
  For ACR 50%, the same calculation is made with 50% improvement, ACR 20%, same calculation with 20% improvement

OTHER OUTCOMES:
Nanostring | At Week 4
  Normalization of inflammatory gene signature

CONTACTS AND LOCATIONS:
Overall Officials: Curdin Conrad, Professor, Principal Investigator — CHUV centre hospitalier universitaire vaudois
Locations (1):
- Centre hospitalier universitaire vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No